CLINICAL TRIAL: NCT03491280
Title: Diagnostic Research in Patients With Rare Diseases - Solving the Unsolved Rare Diseases
Acronym: DiRiP-RD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Prof. Dr. Ludger Schöls, Principal investigator, University Hospital Tuebingen
Other Study IDs: DiRiP-RD
Record Dates: First submitted 2017-12-20; First posted 2018-04-09 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Rare Diseases; Genetic Predisposition
Keywords: Rare Diseases; Genetic Predisposition; Omics Technology; Next Generation Sequencing (NGS)
MeSH Terms: conditions — Rare Diseases; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Subjects with unclear rare diseases, clinically characterized in the context of outpatient/ inpatient standard care at the University Hospital Tübingen (UKT) or cooperating location, genetic diagnostic (NGS diagnostic) must be performed.
  Interventions: Genetic: NGS Diagnostic
- Group 2: Subjects with unclear rare diseases, genetic diagnostic (NGS diagnostic) is already performed.
  Interventions: Genetic: NGS Diagnostic

INTERVENTIONS:
Genetic: NGS Diagnostic — Blood take for genetic diagnostic.
  Other Names: Omics Technology

SUMMARY:
The DiRiP study will enroll patients (n = 3500) with unclear rare diseases and suspected genetic reasons. In group 1 (n = 500) subjects are clinically characterized in the context of outpatient/ inpatient standard care at the UKT or cooperating location, NGS analyzes and other omics analyzes (transcriptomics, proteomics, metabolomics), functional cell biology studies will be performed. In group 2 diagnostics is already performed.

The DiRiP-study fully integrates with the newly formed European Reference Networks (ERNs) for rare diseases, and in particular the ERN-RND, -EURO-NMD, -ITHACA, and -GENTURIS.

DETAILED DESCRIPTION:
In the DiRiP-RD study (monocentric, prospective, open-label diagnostic study), patients with genetically unexplained diseases will be analyzed or re-analyzed from existing datasets for further omics analysis. These are evaluated with regard to the following questions:

Primary:

* Verification of the genetic causes of unclear genetic diseases

Secondary:

* Improve number of diagnoses of unclear syndromes
* Further characterization of the identified gene defects
* Number of patients receiving appropriate therapy after successful diagnosis. In addition, patient phenotype and genotype data can be collected using a software tool for collecting and analyzing phenotypic information of patients with genetic disorders ( PhenoTips®) software to facilitate data exchange within the UKT, with external collaborators and data transfer to the Solve-RD project.

ELIGIBILITY:
Inclusion Criteria:

* Unclear diagnosis
* Suspected genetic cause of the disease

Exclusion Criteria:

* Missing informed consent of the patient/ legal guardian

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study recruit both underage and adult persons (male and female) with unclear genetic syndromes who present themselves for consultation at the UKT and who are suspected of having a genetic cause of the disease.
Sampling Method: Non-Probability Sample
Enrollment: 5500 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Molecular genetic | Day 1
  Verification of the genetic causes of unclear genetic diseases

SECONDARY OUTCOMES:
Number of diagnoses | Day 1
  Improve number of diagnoses of unclear syndromes
Characterization of gene defects | Day 1
  Further characterization of the identified gene defects
Number of patients receiving appropriate therapy after successful diagnosis | Day 1
  Number of patients receiving appropriate therapy after successful diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Holm Graessner, Dr., Study Chair — Managing Director
Locations (1):
- University Hospital, Tübingen, Germany